CLINICAL TRIAL: NCT06389539
Title: A Randomized, Double-Blind, Placebo-Controlled, Clinical Food Trial of Probiotic/Prebiotic Medical Food for the Dietary Management of Age Related Bone Loss
Brief Title: Synbiotic to Attenuate Resorption of the Skeleton
Acronym: STARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: Solarea Bio, Inc (Industry); Beth Israel Deaconess Medical Center (Other); Tufts University (Other); MaineHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Pro00070958
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis; Inflammation; Aging
Keywords: Dietary probiotics; Dietary prebiotics; Gut microbiome; Older women; Randomized Controlled Trial
MeSH Terms: conditions — Osteoporosis; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either SBD111 medical food or placebo capsules for a period of 18 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study staff involved in participants' outcome assessments will be masked to the intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBD111 medical food (Experimental): This group will receive SBD111 medical food capsules to be consumed over 18 months.
  Interventions: Other: SBD111 medical food
- Placebo (Placebo Comparator): This group will receive placebo capsules to be consumed over 18 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: SBD111 medical food — SBD111 medical food is a defined microbial assemblage (DMA) consisting of oligofructose and dried berry powder (prebiotics), a Pseudomonas fluorescens, a Lactobacillus brevis, a Leuconostoc mesenteroides, a Lactobacillus plantarum, and a Pichia kudriavzevii (yeast).
  Arms: SBD111 medical food
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, double blind, placebo controlled clinical trial will test the efficacy of a probiotic/prebiotic combination ("synbiotic") on the skeleton in older women.

DETAILED DESCRIPTION:
There are currently no consistent guidelines on how middle aged and older adults can maintain healthy bone mass as they age. Hence, there is an unmet need for safe and effective dietary interventions for the metabolic processes underlying bone loss. The objective of this project, is to test the efficacy of a probiotic/prebiotic combination or synbiotic i.e. Solarea Bio defined microbial assemblage 111 (SBD111) medical food on the skeleton of older women.

Aim 1: To determine the effect of 18 months of daily intake of SBD111 medical food on the primary outcome of lumbar spine dual energy x-ray absorptiometry (DXA) bone mineral density (BMD) and secondary outcomes (Biomechanical Computed Tomography analysis (BCT)-derived vertebral compressive strength, volumetric BMD (vBMD), and markers of bone turnover) in women.

Hypothesis 1a: BMD, vertebral compressive strength, and vBMD will be greater in women randomized to SBD111 medical food compared to placebo.

Hypothesis 1b: Biochemical markers of bone turnover will decrease with SBD111 medical food use compared to placebo.

Aim 2: To determine the effect of 18 months of daily intake of SBD111 medical food on markers of inflammation and gut microbiome function (secondary outcomes) in women.

Hypothesis 2a: Markers of inflammation [interleukin 17A (IL17A) and tumor necrosis factor alpha (TNF-α)] will be reduced with SBD111 medical food use compared to placebo.

Hypothesis 2b: Functional genes and pathways related to fiber breakdown (glycosyl hydrolases), menaquinone 7 production, and short chain fatty acid (SCFA) production, will be enriched in stool metagenomes and upregulated in stool metatranscriptomes from those receiving SBD111 medical food compared to placebo.

Eligible women will be randomized to SBD111 medical food versus placebo capsules for 18 months. Assessments will be made at the in-person baseline visit, 9-month and 18-month follow-up visits as well as monthly telephone calls.

The primary outcome is lumbar spine BMD (g/cm2) and secondary outcomes include vertebral compressive strength (N), vBMD (g/cm3), and bone biomarkers.

Intent-to-treat analysis will be conducted for all endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provided written informed consent.
* 2. Stated availability throughout entire study period and willingness to fulfill all details of the protocol.
* 3. Age 60 years and above.
* 4. DXA-BMD of the hip and spine (T-score) > -2.5. Women with a BMD T score ≤ -2.5 (i.e. women with low BMD indicating osteoporosis) will also be considered if they have decided not to accept the standard of care use of osteoporosis medications for the entire duration of their participation in the study.
* 5. Women with a history of major low-trauma fragility fractures (hip, forearm, humerus, spine) since the age of 50 years will be considered if they are not currently using osteoporosis medications, or if they have decided not to accept the standard of care osteoporosis medications, even if diagnosed with osteoporosis during the screening procedure.
* 6. Serum 25-hydroxyvitamin D ≥ 20 ng/mL.
* 7. Normal renal function (eGFR >50 ml/min).
* 8. Have chosen to not accept the standard of care use of osteoporosis medications for the duration of the study.
* 9. Willing to comply with protocol and report on compliance and side effects during the study period.

Exclusion Criteria:

* 1. BMI greater than 40 kg/m2.
* 2. Participants consuming dietary supplements (fish oil, probiotics/prebiotics, and fiber) in the prior month, and unwilling to avoid these supplements for the duration of the study.
* 3. Participants using osmotic laxatives >1 per week and unwilling to avoid use for the duration of the study.
* 4. Known or suspected allergies to probiotics, rice, edible fruit extract or berries.
* 5. Antibiotic use in the past 3 months. Participants placed on an antibiotic after enrollment will be retained.
* 6. History of drug and/or alcohol abuse at the time of enrolment.
* 7. Presence of any of the following:
* a. History of other bone disorders (e.g. Paget's disease).
* b. History of moderate to severe scoliosis.
* c. History of cancer other than skin cancer <5 years in remission, autoimmune disease, immune problems such as AIDS, type 1 or 2 diabetes.
* d. History of colon resection, any disease that could interfere with the intestinal barrier function such as ulcerative colitis, irritable bowel syndrome or Crohn's disease or any chronic bowel condition.
* e. Women with untreated hyperparathyroidism.
* f. History of chronic antibiotic use.
* g. History of bariatric surgery.
* h. History of partial colectomy.
* i. History of pancreatic disease.
* j. History of active hepatitis B, hepatitis C, cirrhosis, metabolic dysfunction-associated steatotitc liver disease (MASLD), fatty liver or chronic liver disease.
* k. Current bone marrow disorders such as myelodysplastic syndrome or anemia requiring transfusions.
* l. Abnormalities of the spine determined by the study physician to interfere with the assessment of bone mineral density.
* m. Current smoking or use of nicotine products within the past 6 months.
* n. Current use of marijuana and unwilling to abstain during the study period.
* o. Major abdominal surgery within the last 3 months.
* p. Colonoscopy within the last 1 month.
* q. Colonoscopy planned in the next 18 months and unwilling to reschedule it.
* r. Indwelling catheter, implanted hardware/prosthetic device or feeding tube.
* s. Any medical condition that could interfere with the conduct of the study.
* 8. Treatment with calcitonin, estrogens, selective estrogen receptor modulators, progestins, anabolic steroids, or glucocorticoids in the past 6 months.
* 9. Treatment with bisphosphonates in the past 3 years.
* 10. Previous treatment with parathyroid hormone (PTH), abaloparatide, romosozumab or denosumab in the last year or current coumadin use.
* 11. Current or previous treatment with glucagon-like peptide (GLP-1) receptor agonists in the last one year.
* 12. Participation in other bone, diet, autoimmune, or GI related clinical trials in the last 6 months. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.
* 13. Participants who plan on changing diet and/or exercise regime during trial participation.
* 14. Screening laboratory tests greater than upper normal limit (ULN) or less than lower normal limit (LLN):
* Serum 25-hydroxyvitamin D <20 ng/mL
* Renal dysfunction (eGFR ≤50 ml/min)
* 15. Seated blood pressure greater than equal to 160 mm Hg or seated diastolic blood pressure greater than equal to 100mm Hg.
* 16. Short Blessed Test score >10 or judged by the research staff as unable to follow the study protocol.
* 17. Any other condition that in the opinion of the investigator or study clinician would jeopardize the safety or rights of the volunteer participating in the study or would make it unlikely the volunteer could complete the study.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Lumbar spine BMD (g/cm2) | Change over 18 months
  BMD of the lumbar spine (L1-L4) will be measured at the baseline exam, 9-month, and 18-month final follow-up visit

SECONDARY OUTCOMES:
Vertebral compressive strength (N) | Change over 18 months
  Quantitative computed tomography (QCT) scans acquired at baseline and 18-months will be used to estimate vertebral compressive bone strength using Biomechanical Computed Tomography (BCT, VirtuOst, O.N. Diagnostics, Berkeley, CA).
volumetric BMD | Change over 18 months
  Measurements of integral and vertebral trabecular vBMD at L1-L3.
C-terminal cross-linked telopeptide of type I collagen (β-CTX) | Change over 18 months
  A biochemical marker of bone resorption
Procollagen Type I Intact N-terminal Propeptide (P1NP) | Change over 18 months
  A biochemical marker of bone formation

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Sahni, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew SeniorLife, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT06389539/SAP_000.pdf